CLINICAL TRIAL: NCT06756295
Title: A Phase I/ II Study of Fragmented Autoantigen Stimulated T-cell-immunotherapy Combined with Radiotherapy (FAST-CR)
Acronym: FAST-CR
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fengming Kong (Other)
Collaborators: The University of Hong Kong-Shenzhen Hospital (Other); Peking University (Other)
Responsible Party: Sponsor-Investigator, Fengming Kong, Tenured Clinical Professor, The University of Hong Kong-Shenzhen Hospital
Organization: The University of Hong Kong-Shenzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCOG0052
Record Dates: First submitted 2024-12-31; First posted 2025-01-01 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer, Colorectal Cancer; Melanoma; Lung Cancer
Keywords: tumor vaccine; immunogenic cell death; TCV
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Melanoma; Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard treatment + adjuvant (No Intervention): Patients in the control group include two categories: (1) surgical patients who receive standard postoperative treatment according to guidelines, and (2) non-surgical patients who receive standard RT.
- Standard treatment + individualized tumor FAST vaccine combination (including adjuvant) (Experimental): Surgical Patients: These patients will receive standard postoperative treatment according to guidelines. In Phase I of the trial, they will be randomly administered the aforementioned low, medium, or high doses of the FAST vaccine (P12). In Phase II, the optimal dose will be selected for each patient (as assessed by an expert panel).
  Non-Surgical Patients: Before starting the tumor vaccine, these patients will first undergo three sessions of precision radiotherapy (the doctor will determine whether the patient should receive 2 Gy × 3 or 8 Gy × 3, depending on the patient's condition). After completing the radiotherapy, the individualized tumor vaccine will be administered one week later. Similarly, in Phase I, these patients will receive the low, medium, or high doses of the FAST vaccine (P12) in a randomized manner. In Phase II, the optimal dose will be selected for each patient (as assessed by the expert panel). Tumor vaccine treatment will be administered in cycles of 5
  Interventions: Biological: individualized tumor FAST vaccine combination (including adjuvant)

INTERVENTIONS:
Biological: individualized tumor FAST vaccine combination (including adjuvant) — Using the patient's individual tumor tissue, an autologous FAST (Fragmented Autoantigen Stimulated T-cell Immunotherapy) vaccine is prepared.
  Arms: Standard treatment + individualized tumor FAST vaccine combination (including adjuvant)

SUMMARY:
Evaluation and exploration of the phase I/II clinical safety and efficacy of personalized FAST(Radiation fueled antigens stimulated T-cell immunotherapy )cancer vaccine combined with radiotherapy.

DETAILED DESCRIPTION:
Tumor whole-cell vaccines, as one of the methods for tumor immunotherapy, have become a key focus of numerous preclinical studies. Among these, the latest approaches include cryopreserved silica-based vaccines/aged cell vaccines and genetically engineered vaccines. These vaccines induce immunogenic cell death in tumor cells, thereby reshaping the body's immune tolerance and promoting in-situ immunity (in-situ vaccination). They enhance the diversity of tumor-associated antigens in the draining lymph nodes, increase the recruitment of T cells, and promote tumor recognition and anti-tumor effects. At the same time, whole-cell vaccines retain all potential antigens of the tumor cells, and this integrity increases the likelihood of immune activation and recognition of distal tumors. Additionally, since the vaccine uses the patient's own tumor tissue, it reduces the risk of immune overactivation that might be caused by foreign components. Preclinical studies have found that in a surgical resection model of primary tumors in experimental animals, the FAST vaccine can significantly inhibit the recurrence and metastasis of tumor lesions, remodel the immune microenvironment of colonized organs, achieve systemic clearance of micro-metastases, suppress tumor recurrence and metastatic progression, and prolong the survival of the experimental animals. On the other hand, many advanced cancer patients in the clinic are not amenable to surgical resection, with a high tumor burden. Moreover, the immune response induced by the whole-cell autologous FAST vaccine requires a certain period to develop. Therefore, in our preclinical study, the investigators combined FAST vaccine administration with radiotherapy to control local tumors in experimental animals. The results showed that this approach significantly enhanced both innate and adaptive immunity, inhibited tumor progression and metastasis, and improved the survival rate of the experimental animals.

This study aims to recruit tumor patients who have undergone standard surgical treatment and those with advanced tumors who have failed standard treatment or experienced disease progression (after failure of third-line treatment),Using the patient's individualized tumor tissue, the investigators will prepare the FAST tumor cell vaccine and combine it with precision radiotherapy to conduct safety and efficacy studies on tumor patients who meet the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

- Voluntarily agree to participate in this study. Age: 18-80 years, regardless of gender. Pathological and imaging diagnosis of advanced or recurrent malignant tumors. The patient must have previously received systemic standard treatment that has failed or led to disease progression, with no effective first-line treatment options available for advanced tumors (effective treatment options refer to the latest clinical guidelines published by the "Chinese Society of Clinical Oncology"). Alternatively, the patient may have undergone standard surgical treatment for tumor relapse prevention.

At least one measurable lesion on imaging (excluding patients who have undergone surgical treatment).

Expected survival ≥ 6 months. ECOG (Eastern Cooperative Oncology Group) performance status score of 0-1. No infectious diseases: HIV antibody negative. Normal hematological function: White blood cells ≥ 3000 cells/µL, hemoglobin ≥ 9 g/dL, platelets ≥ 75,000 cells/µL, absolute neutrophil count > 1000 cells/mm³.

Normal renal function: Serum creatinine (Cr) ≤ ULN × 1.5. Normal liver function: Serum ALT/AST levels less than three times the upper limit of normal.

The patient must be willing to sign an informed consent form and able to comply with the treatment plan.

The patient must undergo tumor resection or biopsy (for vaccine preparation) and peripheral blood collection (for efficacy and prognosis evaluation).

Exclusion Criteria:

- Patients who do not have enough tumor resected or puncture tissue for vaccine production.

Patients who have failed third-line therapy, and whose tumor location or type is not suitable for radiotherapy (as evaluated by the expert group).

Patients whose tumor tissue preparation for the vaccine does not meet the efficacy assessment criteria before enrollment (individualized FAST vaccine Elispot test, see Appendix 4 for specific testing protocol).

Patients with a history of bone marrow or stem cell transplantation. Patients currently participating in other therapeutic clinical trials; Traditional Chinese medicine clinical trials.

Patients with active bacterial or fungal infections as per NCI-CTC (National Cancer Institute Common Terminology Criteria for Adverse Events) CTCAE 5.0.

Patients infected with HIV (Human Immunodeficiency Virus), HCV (Hepatitis C Virus), HBV (Hepatitis B Virus), severe asthma, autoimmune diseases, immunodeficiency, or those undergoing immunosuppressive therapy.

Patients with herpesvirus infection (except those whose lesions have scabbed for more than 4 weeks).

Patients with respiratory viral infections (except those who have been cured for more than 4 weeks).

Patients with severe coronary artery or cerebrovascular diseases, or other diseases that the investigator considers should be excluded.

Patients with clinical, psychological, or social factors that affect their ability to provide informed consent for the study.

Patients with a history of autoimmune diseases, such as but not limited to inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Patients with autoimmune-related thyroid diseases and vitiligo are allowed.

Patients with severe chronic or acute comorbidities, such as heart disease (NYHA Class III or IV), liver disease, or other diseases that the principal investigator considers to pose unnecessary high risk in relation to the study drug treatment.

Patients who have a second malignant tumor at the same time (or within the past 5 years), except for melanoma skin cancer, cervical carcinoma in situ, controlled superficial bladder cancer, or other treated carcinoma in situ.

Patients with active acute or chronic infections, including urinary tract infections, HIV (as confirmed by ELISA and Western Blot). HIV-infected individuals may be excluded because immunosuppression could prevent them from responding to the vaccine; chronic hepatitis patients may be excluded due to concerns that vaccination could exacerbate their hepatitis.

Patients with a history of drug or peptide allergies, or allergies to other potential immunotherapies.

Patients undergoing chronic steroid treatment (or other immunosuppressive agents, such as azathioprine or cyclosporine A) will be excluded due to potential immunosuppression. Patients must stop any steroid treatment 6 weeks prior to enrollment (except for drugs used for chemotherapy, contrast-enhanced imaging, or acute treatment of complications such as gout attacks <5 days).

Patients with acute or chronic skin diseases will be excluded, as these conditions could affect the injection into the skin of the limbs or the subsequent evaluation of potential skin reactions.

Patients without legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
safe | one month
  The primary endpoint of this study: The Phase I safety evaluation will involve a 3×3 dose escalation of the vaccine (based on a similar international clinical trial, NCT05366062, with low, medium, and high-dose groups, each group receiving 500,000, 1 million, and 2 million cancer cell fragments, respectively, with 3 participants per group). The safety profile will be summarized, including the incidence and severity of adverse events (Evaluation criteria: Treatment toxicity graded according to CTCAE 5, (Common Terminology Criteria for Adverse Events version 5). If the summary of Phase I toxicity shows no significant higher toxicity compared to existing immunotherapies, the study will proceed to the Phase II efficacy trial.

SECONDARY OUTCOMES:
OS (Overall Survival) | 5 years
  OS (Overall Survival) is defined as the time from the start of FAST treatment to death from any cause.
DFS (disease free survival) | 5 years
  the period of time from the end of treatment or the initial diagnosis of the disease during which the patient shows no signs of disease recurrence, metastasis, or the appearance of new tumors. It is commonly used to assess the disease-free period following cancer treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Chen H, Shen Q, Liu Y, Li P, Ma Y, Wang Y, Li S, Yan X, Liu L, Shuai J, Wu M, Ouyang Q, Kong FS, Yang G. Fragment Autoantigens Stimulated T-Cell-Immunotherapy (FAST) as a Fast Autologous Cancer Vaccine. Adv Sci (Weinh). 2025 Jul;12(26):e2502937. doi: 10.1002/advs.202502937. Epub 2025 Mar 26. PMID 40135850